CLINICAL TRIAL: NCT01934634
Title: Phase I Trial of the Proapoptotic Agonist, LCL161, and Gemcitabine Plus Nab-Paclitaxel in Patients With Metastatic Pancreatic Cancer
Brief Title: Phase I Trial of LCL161 and Gemcitabine Plus Nab-Paclitaxel in Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: US Oncology Research (Industry)
Collaborators: Novartis Pharmaceuticals (Industry); Delta Clinical Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12104; CLCL161AUS03T (Other: Novartis)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Stage IV Pancreatic Cancer; Stage IV metastatic pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — LCL161; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCL161 +Gemcitabine +nab-Paclitaxel (Experimental): LCL161 (tablets): 600, 1200, or 1800 mg once a week (Day 1, 8, 15) for 3 weeks, every 28 days Gemcitabine IV: 1,000 mg/m2 once a week (Day 1, 8, 15) for 3 weeks, every 28 days nab-paclitaxel IV: 100 or 125 mg/m2 once a week (Day 1, 8, 15) for 3 weeks, every 28 days
  Interventions: Drug: LCL161; Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: LCL161 — LCL161 (tablets): 300, 600, 1200, or 1800 mg once a week (Day 1, 8, 15) for 3 weeks, every 28 days
Drug: Gemcitabine — Gemcitabine IV: 1,000 mg/m2 once a week (Day 1, 8, 15) for 3 weeks, every 28 days
  Other Names: Gemzar
Drug: nab-Paclitaxel — nab-paclitaxel IV: 125 mg/m2 once a week (Day 1, 8, 15) for 3 weeks, every 28 days
  Other Names: Abraxane

SUMMARY:
The goal of this study is to identify the maximum tolerated dose and dose-limiting side effects of LCL161 in combination with gemcitabine and nab-paclitaxel and to provide safety data in patients with measurable metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Improved therapeutic options for advanced pancreatic adenocarcinoma treatment need to continue to be investigated. Since 1997, gemcitabine has been the agent of choice for first-line therapy in advanced pancreatic cancer, with a median survival of 5.7 months, and a 20% 1-year survival (Eli Lilly 1996). Combination therapies using gemcitabine as a backbone have been investigated, but none are superior to gemcitabine monotherapy, except for a modest increase in overall survival (OS) with erlotinib and gemcitabine (Moore et al 2007). In a study of FOLFIRINOX compared with gemcitabine as first-line therapy in 342 metastatic pancreatic cancer patients, median OS was 11.1 months in the FOLFIRINOX group and 6.8 months in the gemcitabine group; however, the FOLFIRINOX group experienced more adverse events particularly febrile neutropenia (Conroy et al 2011).

LCL161 is a biostable, cell-permeable, small molecular weight Smac-mimetic compound. It is an orally bioavailable pan-IAP inhibitor that demonstrates anti-tumor efficacy as a single agent in a small subset of cell lines, and in many more cell lines and xenograft models when given in combination with paclitaxel.

Nanoparticle albumin-bound paclitaxel (nab-paclitaxel) is a formulation that is readily soluble in saline, eliminating the need for lipid-based solvents (ie, Cremophor EL) and corticosteroid and antihistamine premedications for hypersensitivity reactions required for traditional unbound paclitaxel. nab-paclitaxel has also been shown to actively bind to secreted protein acidic and rich in cysteine (SPARC) in the tumor stroma, which is highly expressed in pancreatic cancer and actively binds to the albumin in nab-paclitaxel and further concentrates the drug into the tumor. SPARC expression in the stroma of tumor cells has been associated with poor survival. In a Phase I/II trial (Von Hoff et al 2011) involving 67 patients with metastatic pancreatic adenocarcinoma, the regimen of nab-paclitaxel plus gemcitabine had tolerable adverse effects with substantial antitumor activity, warranting Phase III evaluation.

The Phase III study (MPACT) was a large, international study that determined that survival with nab-paclitaxel plus gemcitabine is superior to gemcitabine alone. nab-paclitaxel plus gemcitabine is a new standard for treatment of patients with metastatic pancreatic cancer (Von Hoff et al 2013). However, although this study shows promise for substantially improving OS in patients with pancreatic adenocarcinoma, insensitivity to these agents is likely to occur due to resistance to apoptosis, which has been observed in laboratory studies to occur for most of the cytotoxic agents used to treat pancreatic cancer in the past (Westphal and Kaltoff 2003). Exploitation of the apoptosis pathway may ultimately provide more effective, less toxic anticancer therapy that selectively circumvents treatment-resistant pathways.

Based on the above, there is a high likelihood that LCL161 in combination with nab-paclitaxel and gemcitabine will be determined to be safe and well tolerated, and will show substantial antitumor activity, warranting Phase II evaluation.

Up to 24 patients will be enrolled in Part A - Phase I Safety study. If the combination therapy is determined to be safe and well tolerated and shows substantial antitumor activity, a safety expansion cohort of 12 additional patients will be enrolled in Part B - Efficacy study to further confirm the tolerability and efficacy of LCL161 with an endpoint of complete response (CR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to any screening procedures.
2. A signed Patient Authorization Form (HIPPA) has been obtained prior to registration.
3. Age 18 years or older.
4. Willing and able to comply with scheduled visits, treatment plan and laboratory tests
5. Patient is able to swallow and retain oral medication.
6. Histologically or cytologically documented measureable metastatic (Stage IV) pancreatic cancer with disease by computed tomography scan as defined by RECIST Version 1.1.
7. ECOG performance status 0-1.
8. Required baseline laboratory status:

   * Hemoglobin (Hgb) ≥ 90 g/L (9 g/dL)
   * Platelets ≥ 100 x 109/L (100,000/mm3)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/mm3)
   * Serum total bilirubin ≤ 1.5 x ULN (upper limit of normal)
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN, except for patients with tumor involvement of the liver who must have AST and ALT ≤ 5 x ULN
   * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 40 mL/min
9. Patient did not receive previous treatment for Stage IV pancreatic cancer. Note: However, prior adjuvant treatment with fluorouracil or gemcitabine administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed. If patient received adjuvant therapy, tumor recurrence must have occurred ≥ 6 months after the last treatment.

Exclusion Criteria:

1. Patient has any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while on the study or that could confound discrimination between disease- and study treatment-related toxicities.
2. Patient has impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * History or presence of ventricular tachyarrhythmia
   * Presence of unstable atrial fibrillation (ventricular response > 100 bpm); Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria
3. Patient is currently receiving chronic (> 14 days) treatment with corticosteroids at a dose ≥ 10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug.
4. Patient is currently receiving treatment with agents that are metabolized solely through CYP3A4/5 and have a narrow therapeutic index or are strong CYP2C8 inhibitors; or are receiving treatment with agents that carry a risk for QT prolongation and are CYP3A substrates. Caution should be used in patients taking other CYP2C8- or CYP3A4/5-interacting agents.
5. Patient has impairment of Gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LCL161.
6. Patient is a pregnant or breast feeding (lactating) woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive β-HCG laboratory test (> 5 mIU/mL).
7. Patient is a woman of child-bearing potential, defined as all women physiologically capable of becoming pregnant and refusing to use highly effective methods of contraception during dosing and for 90 days after study treatment. Highly effective contraception methods include:

   * Total abstinence or
   * Male partner or female sterilization or
   * Combination of any 2 of the following (a+b or a+c, or b+c):

     1. Use of oral, injected, or implanted hormonal methods of contraception
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
     3. Barrier methods of contraception: condom for male partner or occlusive cap (diaphragm or cervical/vault caps) with spermicidal form/gel/film/cream/ vaginal suppository.

   Note: Postmenopausal women are allowed to participate in this study. Women are considered postmenopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (eg, age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks earlier. In the case of oophorectomy alone, a woman is considered to be not of child bearing potential only when her reproductive status has been confirmed by follow-up hormone level assessment.
8. Patient is abstaining from using a condom. Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
9. Patient has a history of lymphoma with or without treatment.
10. Patient has a history of interstitial pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of LCL161 | 1.6 years
  The maximum dose of LCL161 (tablets: 600, 1200, or 1800 mg once a week (Day 1, 8, 15) for 3 weeks, every 28 days) that is tolerated by the patients.
Percentage of patients with Dose-Limiting Toxicities | 1.6 years
  The percentage of patients that have side effects that require dosage of LCL161 to be stopped or reduced.

SECONDARY OUTCOMES:
Objective Response Rate | 1.6 years
  Number of patients with Complete Response or Partial Response

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M. Coyle, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health; Carlos H. Becerra, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 2 Sites, Incl Tyler, TX and Dallas, TX, Texas, United States